CLINICAL TRIAL: NCT03222336
Title: Study of Natural History Among Patients With Chinese Hotspot Late-onset Fabry Mutation IVS4+919G>A Through Family Pedigree Analysis
Brief Title: Natural History in Fabry Patients With IVS4+919G>A Mutation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, vghtpe user, Director, Pediatric Genetic and Endocrinology Division, Taipei Veterans General Hospital, Taiwan
Other Study IDs: Fabry Version 1.0 VGHTP 2016
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Fabry Disease, Cardiac Variant
MeSH Terms: conditions — Fabry Disease, Cardiac Variant | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Family pedigree and data collection — 1. Enroll first generation (newborn), at least one member from second (parent) and third generation (grandparent) for a complete IVS4 family tree mapping.
  2. Collect and analyze medical history, genetic and biochemical assessment data

SUMMARY:
Fabry disease is caused by the deficiency or absence of alpha-galactosidase A (α-Gal A) activity, leading to progressive deposition of glycosphingolipids, mainly globotriaosylceramide (Gb3), in the lysosomes of multiple tissues and organs. In Taiwan, Dr. Niu first revealed a surprisingly high incidence (approximately one in 1,600 males) of a cardiac variant GLA splicing mutation, IVS4+919G>A, in newborn screening. Patients who carried the IVS4 + 919G > A mutation and were older than 40 years had a higher prevalence of hypertrophic cardiomyopathy. Endocardial biopsy of these patients with hypertrophic cardiomyopathy showed significant Gb3 accumulation in the cardiomyocytes. Although the hotspot IVS4+919G>A mutation is now being observed with greater frequency, understanding of the natural course of cardiac variant Fabry disease with this specific mutation remains limited. Therefore, our study would like to conduct a study to approach the natural history among patients with Chinese hotspot late-onset Fabry mutation IVS4+919G>A through family pedigree analysis.

DETAILED DESCRIPTION:
Fabry disease is caused by the deficiency or absence of alpha-galactosidase A (α-Gal A) activity, leading to progressive deposition of glycosphingolipids, mainly globotriaosylceramide (Gb3), in the lysosomes of multiple tissues and organs. The frequency of classic Fabry disease has been estimated as one in 40,000, and its symptoms typically manifest during childhood, including acroparesthesias, angiokeratoma, corneal opacities, and anhidrosis (Desnick et al. 2001; Ries et al. 2005). Originally thought to be less severe in females (Desnick et al. 2001), more recent evidence indicates that symptoms of this X-linked disorder can manifest as severely in females as in males (Mehta et al. 2004; Wilcox et al. 2008), although they generally occur later in life and show greater variation in severity among female patients (Deegan et al. 2006).

Atypical, late-onset phenotypes have been reported that lack these classic symptoms but instead present with cardiac (Nakao et al. 1995), renal (Nakao et al. 2003), or cerebrovascular disease (Brouns et al. 2010). The frequency of atypical Fabry disease is unknown, but it has been suggested to be more common than previously believed (Nakao et al. 1995). In Taiwan, Dr. Niu first revealed a surprisingly high incidence (approximately one in 1,600 males) of a cardiac variant GLA splicing mutation, IVS4+919G>A, in newborn screening (Chong et al. 2008). Affected males with IVS4+919G>A mutation typically lack the angiokeratomas, acroparesthesias, hypohidrosis, gastrointestinal abnormalities and corneal opacities that are characteristic of the classic, early-onset, more severe phenotype and may manifest cardiac disease with LVH leading to HCM in the third to sixth decades of life (Desnick et al. 2001, von Scheidt W, et al. 1991, Nakao et al. 1995, Nakao et al. 2003). In Dr. Niu's study, patients who carried the IVS4 + 919G > A mutation and were older than 40 years had a higher prevalence of hypertrophic cardiomyopathy (72% of males and 35% of females) (Tai et al., 2012). Endocardial biopsy of these patients with hypertrophic cardiomyopathy showed significant Gb3 accumulation in the cardiomyocytes which is the typical pathological change in patient with classical Fabry disease. Lin et al's previous study (Lin et al. 2010) showed that a high proportion of adults (>40 years of age) carrying the IVS4 +919G>A mutation experienced microalbuminuria and retinal vessel tortuosity, but symptoms involving these organs were very mild and did not cause significant morbidity. Although the hotspot IVS4+919G>A mutation is now being observed with greater frequency, understanding of the natural course of cardiac variant Fabry disease with this specific mutation remains limited.

Primary objective :

* To map the IVS4 family tree and identify obligate carriers with Chinese hotspot late-onset Fabry mutation IVS4+919G>A through pedigree analysis.
* To explore and enhance the understanding of the clinical manifestation, disease severity and natural history of patient with Chinese hotspot late-onset Fabry mutation IVS4+919G>A in Taiwan.

Primary End Point :

- Completeness of IVS4 family tree mapping and obligate carrier identification within their family pedigree.

Definition of family tree completeness:

- Enroll first generation (newborn), at least one member from second (parent) and third generation (grandparent) for a complete IVS4 family tree mapping.

Secondary endpoint :

- Collect and analyze medical history, genetic and biochemical assessment data. Perform eGFR and albumin to creatinine ratio (ACR) measurement for renal function assessment, Perform echocardiography and electrocardiography for cardiac function assessment.

ELIGIBILITY:
Inclusion Criteria:

* Fabry IVS4 female newborn family members.
* Patients and/or their legal representatives who are willing to provide written informed consent

Exclusion Criteria:

* No blood relatives to the IVS4 female newborn family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective family screening study aim to enrol family members from pre-identified IVS4 female newborn's family. IVS4 female newborn's family member will be invited to join the family screening study with written informed consent prior to any specific study procedure. After written informed consent process, a series of screening examination will be conducted at screening visit which included medical history interview, physical examination, α-Gal A enzyme activity test, genetic test, plasma lyso-GB3, renal function and cardiac function assessment as well as pedigree data analysis for IVS4 family tree mapping.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Completeness of IVS4 family tree mapping and obligate carrier identification within their family pedigree | First patient in : 30-Sep-2017; Last Patient out : 1-June-2020

REFERENCES:
- [Background] Brouns R, Thijs V, Eyskens F, Van den Broeck M, Belachew S, Van Broeckhoven C, Redondo P, Hemelsoet D, Fumal A, Jeangette S, Verslegers W, Baker R, Hughes D, De Deyn PP; BeFaS Investigators. Belgian Fabry study: prevalence of Fabry disease in a cohort of 1000 young patients with cerebrovascular disease. Stroke. 2010 May;41(5):863-8. doi: 10.1161/STROKEAHA.110.579409. Epub 2010 Apr 1. PMID 20360539
- [Background] Chong KW, Lu YH, Hsu JH, Lo MY, Hsiao CY, Niu DM (2008) High incidence of cardiac variant of Fabry disease in Taiwanese revealed by newborn screening Conference High incidence of cardiac variant of Fabry disease in Taiwanese revealed by newborn screening, Hualien, Taiwan, 2008, pp 92-98
- [Background] Deegan PB, Baehner AF, Barba Romero MA, Hughes DA, Kampmann C, Beck M; European FOS Investigators. Natural history of Fabry disease in females in the Fabry Outcome Survey. J Med Genet. 2006 Apr;43(4):347-52. doi: 10.1136/jmg.2005.036327. Epub 2005 Oct 14. PMID 16227523
- [Background] Desnick RJ, Ioannou YA, Eng CM (2001) a-Galactosidase A deficiency: Fabry disease. In: Scriver CR, Beaudet AL, Sly WS, Valle D (eds) The metabolic and molecular bases of inherited disease. McGraw-Hill, New York, pp 3733-3774
- [Background] Lin HY, Huang CH, Yu HC, Chong KW, Hsu JH, Lee PC, Cheng KH, Chiang CC, Ho HJ, Lin SP, Chen SJ, Lin PK, Niu DM. Enzyme assay and clinical assessment in subjects with a Chinese hotspot late-onset Fabry mutation (IVS4 + 919G-->A). J Inherit Metab Dis. 2010 Oct;33(5):619-24. doi: 10.1007/s10545-010-9166-7. Epub 2010 Sep 7. PMID 20821055
- [Background] Mehta A, Ricci R, Widmer U, Dehout F, Garcia de Lorenzo A, Kampmann C, Linhart A, Sunder-Plassmann G, Ries M, Beck M. Fabry disease defined: baseline clinical manifestations of 366 patients in the Fabry Outcome Survey. Eur J Clin Invest. 2004 Mar;34(3):236-42. doi: 10.1111/j.1365-2362.2004.01309.x. PMID 15025684
- [Background] Nakao S, Takenaka T, Maeda M, Kodama C, Tanaka A, Tahara M, Yoshida A, Kuriyama M, Hayashibe H, Sakuraba H, et al. An atypical variant of Fabry's disease in men with left ventricular hypertrophy. N Engl J Med. 1995 Aug 3;333(5):288-93. doi: 10.1056/NEJM199508033330504. PMID 7596372
- [Background] Nakao S, Kodama C, Takenaka T, Tanaka A, Yasumoto Y, Yoshida A, Kanzaki T, Enriquez AL, Eng CM, Tanaka H, Tei C, Desnick RJ. Fabry disease: detection of undiagnosed hemodialysis patients and identification of a "renal variant" phenotype. Kidney Int. 2003 Sep;64(3):801-7. doi: 10.1046/j.1523-1755.2003.00160.x. PMID 12911529
- [Background] Ries M, Gupta S, Moore DF, Sachdev V, Quirk JM, Murray GJ, Rosing DR, Robinson C, Schaefer E, Gal A, Dambrosia JM, Garman SC, Brady RO, Schiffmann R. Pediatric Fabry disease. Pediatrics. 2005 Mar;115(3):e344-55. doi: 10.1542/peds.2004-1678. Epub 2005 Feb 15. PMID 15713906
- [Background] von Scheidt W, Eng CM, Fitzmaurice TF, Erdmann E, Hubner G, Olsen EG, Christomanou H, Kandolf R, Bishop DF, Desnick RJ. An atypical variant of Fabry's disease with manifestations confined to the myocardium. N Engl J Med. 1991 Feb 7;324(6):395-9. doi: 10.1056/NEJM199102073240607. No abstract available. PMID 1846223
- [Background] Tai CL, Liu MY, Yu HC, Chiang CC, Chiang H, Suen JH, Kao SM, Huang YH, Wu TJ, Yang CF, Tsai FC, Lin CY, Chang JG, Chen HD, Niu DM. The use of high resolution melting analysis to detect Fabry mutations in heterozygous females via dry bloodspots. Clin Chim Acta. 2012 Feb 18;413(3-4):422-7. doi: 10.1016/j.cca.2011.10.023. Epub 2011 Oct 29. PMID 22063097
- [Background] Wilcox WR, Oliveira JP, Hopkin RJ, Ortiz A, Banikazemi M, Feldt-Rasmussen U, Sims K, Waldek S, Pastores GM, Lee P, Eng CM, Marodi L, Stanford KE, Breunig F, Wanner C, Warnock DG, Lemay RM, Germain DP; Fabry Registry. Females with Fabry disease frequently have major organ involvement: lessons from the Fabry Registry. Mol Genet Metab. 2008 Feb;93(2):112-28. doi: 10.1016/j.ymgme.2007.09.013. Epub 2007 Nov 26. PMID 18037317